CLINICAL TRIAL: NCT01440608
Title: Randomized, Double-blind, Placebo-controlled Trial Evaluating the Impact of High-dose Zinc Therapy and Albendazole in the Treatment of Sub-clinical Environmental Enteropathy in Rural Malawian Children
Brief Title: Effectiveness of High-dose Zinc Therapy and Albendazole in the Treatment of Environmental Enteropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJM-zincalbendazole
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Enteropathy
MeSH Terms: conditions — Intestinal Diseases | interventions — Albendazole; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Zinc therapy (Experimental): High-dose zinc, equivalent 20 mg elemental zinc, to be given once per day for 14 days
  Interventions: Dietary Supplement: High-dose Zinc
- Albendazole (Experimental): Albendazole to be given once on the day of enrollment. Placebo will then be given for 13 days following.
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Placebo will be given for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Pill form, to be given once, 200 mg dosage for children 1-2 years of age, 400 mg dosage for children 2-3 years of age
  Arms: Albendazole
Drug: Placebo — Pill form, 400 mg dose to be given once per day for 14 days in Placebo arm and 13 days in Albendazole arm following one dose of Albendazole.
  Arms: Placebo
Dietary Supplement: High-dose Zinc — Pill form, equivalent to 20 mg elemental zinc, to be given once per day for 14 days
  Arms: Zinc therapy

SUMMARY:
The purpose of this study is to investigate the therapeutic effectiveness of high-dose zinc therapy and de-worming albendazole as separate interventions in restoring normal gut absorptive and immunological function as measured by the dual sugar permeability test and additional biomarkers in 1-3 year old rural Malawian children at high risk for Environmental Enteropathy.

ELIGIBILITY:
Inclusion Criteria:

* 1-3 years of age
* Lives in study villages

Exclusion Criteria:

* Unable to drink 100 mL of sugar water
* Demonstrating evidence of severe acute malnutrition, WHZ < or = -3, presence of bi-pedal pitting edema
* Apparent need for acute medical treatment for an illness or injury
* Parent refusal to participate and return for 7-week follow-up

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in urine lactulose:mannitol (L:M) ratio following therapy course. | 4 weeks, 7 weeks

SECONDARY OUTCOMES:
Change in blood endoCAb | 7 weeks
Change in fecal calprotectin mRNA | 4 weeks, 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Saint Louis Nutrition Project, Blantyre, Malawi

REFERENCES:
- [Derived] Ryan KN, Stephenson KB, Trehan I, Shulman RJ, Thakwalakwa C, Murray E, Maleta K, Manary MJ. Zinc or albendazole attenuates the progression of environmental enteropathy: a randomized controlled trial. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1507-13.e1. doi: 10.1016/j.cgh.2014.01.024. Epub 2014 Jan 22. PMID 24462483